CLINICAL TRIAL: NCT04087369
Title: An Integrated Intervention for Chronic Care Management in Rural Nepal: a Type 2 Hybrid Effectiveness-implementation Study
Brief Title: Integrated NCD Intervention in Rural Nepal
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: This study was withdrawn prior to participant enrollment due to a lack of external funding, dedicated resources, and shifting organizational priorities among research collaborators
Sponsor: Possible (Other)
Collaborators: Nyaya Health Nepal (Unknown); Ministry of Health and Population, Nepal (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: NCDnyaya
Record Dates: First submitted 2019-09-06; First posted 2019-09-12 (Actual); Last update posted 2021-06-25 (Actual); Status verified 2021-06

CONDITIONS: Noncommunicable Diseases; Hypertension; Chronic Obstructive Pulmonary Disease; Diabetes Mellitus, Type 2
Keywords: implementation research; low- and middle-income countries; Nepal; Package of Essential Noncommunicable disease interventions for primary care in low-resource settings; task-shifting; non-physician health workers; digital tools; motivational interviewing
MeSH Terms: conditions — Noncommunicable Diseases; Hypertension; Pulmonary Disease, Chronic Obstructive; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bundled NCD WHO PEN Intervention (Experimental): Mixed-methods type 2 hybrid effectiveness-implementation study to evaluate an integrated NCD care management intervention
  Interventions: Other: Bundled NCD WHO PEN Intervention

INTERVENTIONS:
Other: Bundled NCD WHO PEN Intervention — In the intervention includes the planned roll-out of the World Health Organization's Package of essential noncommunicable disease interventions (WHO PEN) for primary care in low resource settings by the Government of Nepal, Ministry of Health and Population. In addition, this intervention will include three evidence-based components: 1) non-communicable disease (NCD) care integration using mid-level practitioners (MLPs) and community healthcare workers (CHWs); 2) clinical decision support (CDS) tools to ensure quality care in accordance with best practices; and 3) training and supervision of MLPs to provide motivational interviewing (MI) techniques for modifiable risk factor optimization, with a specific focus on tobacco and alcohol use.

SUMMARY:
We will test an NCD intervention bundle incorporating the World Health Organisation (WHO)'s Package for Essential Non-Communicable Disease Interventions (PEN) within an approximate population of 300,000 people in rural Nepal. This intervention integrates three evidence-based approaches for both facility- and community-based NCD care focused on the key areas of Clinical Practice, Counseling, and Technology for two tiers of non-physician healthcare worker - Mid-Level Providers and Community Health Workers: 1) Task-shifting of evidence-based medicine algorithms and clinical skills from PEN protocols to non-physician healthcare workers; 2) Delivering quality counseling based on the Motivational Interviewing Model to drive behavior change with respect to both treatment adherence (defined as medication adherence and follow-up completion) and risk factor modification (alcohol, tobacco, diet, physical activity); 3) Employing a facility- and community-based clinical decision support tool for effective integration of PEN protocols into non-physician healthcare worker workflow. This five-year study will initial test the acceptability and feasibility of the intervention (two years) followed by a type 2 hybrid effectiveness-implementation research trial (three years) to which we will apply the RE-AIM implementation evaluative framework of both outcomes and process indicators. Co-primary outcomes for the intervention bundle will be: a) disease-specific, evidence-based control metrics that measures clinical efficacy; b) qualitative evaluation of acceptability and feasibility that incorporates perspectives of patients, providers, and government stakeholders; and c) an implementation checklist of key intervention process measures.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients aged 18 or older that screen into Nyaya Health Nepal/Possible's chronic disease program for the following conditions: Hypertension, Type II Diabetes Mellitus, COPD, and Asthma OR
2. Adult patients aged 18 or older with end-organ pathology resulting from the aforementioned conditions including the following: Chronic Kidney Disease, Ischemic Heart Disease, Cerebrovascular Disease AND
3. Healthcare staff; mid-level providers serving at district/primary health center-level facility; community health workers serving village clusters, Nyaya Health Nepal/Possible and Government of Nepal/Ministry of Health and Population employees involved in study design, program implementation, data collection, or data analysis processes.

   * Note, study populations 1 and 2 must reside in either Achham or Dolakha (Nepal) districts.

     * Patients must have a noncommunicable note in electronic medical record system at least twice (indicating at least one follow-up visit) and must have minimum 12 weeks in between baseline/endline clinical measures (indicating patients have been followed up for at least 3 months and have 3 months of exposure to intervention).

       * Patients do not need to have been in study for all 3 years. Duration of exposure to intervention will depend on stepped implementation design.

Patients may be identified at Bayalpata Hospital (Achham, Nepal) or Charikot Primary Health Center (Dolakha, Nepal) by facility clinicians. Community health workers can also identify hypertensive patients and refer them to the facility for diagnosis confirmation. Patient enrollment will not be restricted by economic status or caste. Patients will not be recruited exclusively to participate in the study but will undergo routine evaluations, entering the final diagnosis in electronic health record system, tracking progress at each patient contact, the frequency for which is determined by the clinician's recommendation per World Health Organization Package of Essential Noncommunicable disease intervention protocols and the patient's availability. Patients will receive longitudinal care via the community health workers at their homes and at the hospitals by mid-level providers and staff physicians. Their receipt of care is not contingent upon their enrollment in the study; they receive care per routine service delivery.

Exclusion Criteria:

1. Patients migrate from the study are before completion of any of the Package of Essential Noncommunicable disease interventions
2. Patients explicitly request exclusion from the study and decline to consent to the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2023-03 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Type II diabetes mellitus control measure | 24 months
  Percentage of enrolled type II diabetes patients achieving "at goal" status, at the completion of the study period (type II diabetes mellitus: Hemoglobin A1c < 7.5 OR fasting blood sugar <130 mg/dL)
Hypertension control measure | 24 months
  Percentage of enrolled hypertension patients achieving "at goal" status, at the completion of the study period (hypertension: blood pressure <130/80mm Hg or patient-tailored goal per risk stratification)
COPD control measure | 24 months
  Percentage of enrolled COPD patients achieving "at goal" status, at the completion of the study period (COPD: exacerbation status ≤1/3 Anthonisen criteria)

SECONDARY OUTCOMES:
Tobacco use | 24 months
  Percentage of enrolled NCD patients who were using tobacco at enrollment who are non-users or who have reduced by >50% their tobacco intake, at the completion of the study period
Alcohol use | 24 months
  Percentage of enrolled NCD patients who were alcohol drinkers at enrollment who are non-drinkers or who have reduced by >50% alcohol intake, at the completion of the study period

OTHER OUTCOMES:
Home visit coverage (Reach) | 1 month
  Percentage of enrolled NCD patients having a CHW home visit
Clinic visit coverage (Reach) | 1 month
  Percentage of enrolled NCD patients having an MLP visit at the clinic, measured monthly according to the patients indicated to be seen that month based on protocol-based guidelines
Demographic, geographic barriers and facilitators | 24 months
  Percentage of enrolled NCD patients whose CHW has GPS-mapped their households, describing barriers/facilitators to individuals' access, and identifying contributors to variation/inequities
Loss to follow-up (Reach) | 24 months
  Percentage of patients, stratified by demographic data and NCD conditions, that are lost-to-follow-up after enrollment
Monthly patient touch-points (Effectiveness) | 1 month
  Number of monthly per-patient touch-points, including interactions by both MLPs and CHWs
Evidence-based hypertension management (Effectiveness) | 3 months
  Percentage of enrolled hypertension patients in accordance with evidence-based recommendations, as prescribed by clinical algorithms, assessed quarterly by EHR audits
Evidence-based diabetes management (Effectiveness) | 3 months
  Percentage of enrolled diabetes patients in accordance with evidence-based recommendations, as prescribed by clinical algorithms, assessed quarterly by EHR audits
Evidence-based COPD management (Effectiveness) | 3 months
  Percentage of enrolled COPD patients in accordance with evidence-based recommendations, as prescribed by clinical algorithms, assessed quarterly by EHR audits
Village cluster adoption (Adoption) | 24 months
  Percentage of intended village clusters receiving intervention
Timely adoption (Adoption) | 24 months
  Percentage of intended village clusters rolling-out intervention within 3 months of schedule, according to local governance decisions to roll-out the intervention
CHW training adoption (Adoption) | 6 months
  Percentage of CHWs trained in intervention implementation within first six months
CHW retention adoption (Adoption) | 24 months
  Percentage of of trained CHWs retained in their positions at the completion of the study period
MLP training adoption (Adoption) | 24 months
  Percentage of MLPs trained in intervention implementation
MLP retention adoption (Adoption) | 24 months
  Percentage of of trained MLPs retained in their positions at the completion of the study period
Care integration (Implementation) | 1 month
  Percentage of all NCD patients enrolled at the facilities seen by CHWs at home within first month
CHW supervision completion (Implementation) | 3 months
  Percentage of scheduled CHW supervision field visits completed, stratified by CHN and district
CHW supervision review meeting completion (Implementation) | 3 months
  Percentage of scheduled quarterly data review meetings held with CHWs and CHNs
CHW home visit completion (Implementation) | 3 months
  Percentage of enrolled NCD patients with 100% of algorithm-indicated home visits received
CHW home visit fidelity (Implementation) | 3 months
  Percentage of of topics included at each session as dictated by the condition-specific algorithms, assessed during the CHW supervision field visits by CHNs
Referral fidelity (Implementation) | 3 months
  Percentage of patients appropriately referred to MLP care as indicated by the clinical algorithms, assessed during the CHW supervision field visits by CHNs
Referral completion (Implementation) | 3 months
  Percentage of % of patients referred by CHWs seen by MLPs within the prescribed time window according to the clinical algorithms (e.g. 24hours, 72 hours, 1 week)
MLP supervision model (Implementation) | 3 months
  Percentage of enrolled NCD patients appropriately referred to see a physician by MLPs as indicated by the clinical algorithms, assessed during monthly physician supervision sessions
MLP visit fidelity (Implementation) | 1 month
  Percentage of of enrolled NCD patients with 100% of algorithm-indicated facility visits received, assessed during monthly physician supervision sessions
Total intervention cost (Maintenance) | 24 months
  Cost of each intervention component and total costs using the Joint Learning Network costing methodology
Intervention initiation costs (Maintenance) | 24 months
  Percentage breakdown of initial (one-time) costs for intervention (training, equipment, etc)
Intervention maintenance costs (Maintenance) | 24 months
  Percentage breakdown of maintenance (recurring) costs (on-going training, personnel, materials, and other)
Facility vs. community costs (Maintenance) | 24 months
  Percentage of costs of health care divided between facility level and community level
Geographic cost variation (Maintenance) | 24 months
  Variance in costs between village clusters and districts within the intervention catchment area
Out-of-pocket patient costs (Maintenance) | 24 months
  Percentage of costs of health care divided between facility level and community level
Integrated intervention cost-effectiveness analysis (Maintenance) | 24 months
  Pre/post intervention marginal effectiveness for primary outcomes
Cost per unit patient (Maintenance) | 24 months
  Intervention cost per enrolled patient
Cost per capita (Maintenance) | 24 months
  Intervention cost per capita
Projected scale cost(Maintenance) | 24 months
  Projected cost to scale intervention nationally

CONTACTS AND LOCATIONS:
Overall Officials: Sabitri Sapkota, PhD, MPH, Study Director — Possible/Nyaya Health Nepal
Locations (2):
- Nepal (2):
  - Bayalpata Hospital, Sanfebagar-10, Achham/Province 7
  - Charikot Primary Health Center, Chari̇̄koṭ, Dolakha/Province 3

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schwarz D, Dhungana S, Kumar A, Acharya B, Agrawal P, Aryal A, Baum A, Choudhury N, Citrin D, Dangal B, Dhimal M, Gauchan B, Gupta T, Halliday S, Karmacharya B, Kishore S, Koirala B, Kshatriya U, Levine E, Maru S, Rimal P, Sapkota S, Schwarz R, Shrestha A, Thapa A, Maru D. An integrated intervention for chronic care management in rural Nepal: protocol of a type 2 hybrid effectiveness-implementation study. Trials. 2020 Jan 29;21(1):119. doi: 10.1186/s13063-020-4063-3. PMID 31996250